CLINICAL TRIAL: NCT06986668
Title: Comparison of the Efficacy of Paraffin Bath and Peloidotherapy in Patients With Carpal Tunnel Syndrome
Brief Title: Efficacy of Paraffin Bath and Peloidotherapy in Carpal Tunnel Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ümmü Habibe Sarı, MD, Konya Beyhekim Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KonyaBeyhekimTRH9188
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome (CTS); Peloidotherapy; Paraffin Bath; Exercise
Keywords: carpal tunnel syndrome (CTS); Peloidotherapy; paraffin bath; exercise; ultrasound; pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: single-blind, randomized, prospective
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peloidotherapy (Experimental): This group will consist of patients who have received peloid therapy for a total of 15 sessions of 20 minutes at 45 degrees for 3 weeks, 5 days a week, along with a home exercise program.
  Interventions: Other: Peloidotherapy; Other: home exersize
- paraffin bath (Experimental): This group will consist of patients who have received paraffin bath for a total of 15 sessions of 20 minutes for 3 weeks, 5 days a week, along with a home exercise program.
  Interventions: Other: paraffin bath; Other: home exersize
- Home exercise (Experimental): This group will consist of patients who have only been given a home exercise program. Flexor tendon gliding exercises, median nerve gliding exercises, and isometric wrist strengthening exercises will be given as exercises.
  Interventions: Other: home exersize

INTERVENTIONS:
Other: Peloidotherapy — Peloidotherapy stands out among superficial heating physical therapy modalities with its mineral and natural origin.
  Arms: Peloidotherapy
Other: paraffin bath — It is an effective treatment for the treatment of patients' hands, arms and feet by applying the brushing method to different body parts, relieving pain and improving function, thus providing freedom of life.
  Arms: paraffin bath
Other: home exersize — Flexor tendon gliding exercises, median nerve gliding exercises, and isometric wrist strengthening exercises will be given as exercises.

SUMMARY:
Patients diagnosed with mild and moderate idiopathic CTS will be randomly divided into three groups. Patients who received 15 sessions of peloid therapy along with a home exercise program will constitute the first group. The second group will consist of patients who receive 15 sessions of paraffin bath and a home exercise program. Patients who were given only a home exercise program will be included in the third group. "Patients will be evaluated in detail in terms of clinical examination and outcomes three weeks after the end of treatment and again at three months.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compression neuropathy caused by entrapment of the median nerve in the carpal tunnel. There are 2 methods for the treatment of CTS: conservative and surgical. Conservative treatment is mostly applied in patients with mild and moderate CTS. In this study, we aim to evaluate the efficacy of peloid therapy and kinesiobanding technique, which are conservative treatment methods. Patients will be evaluated in terms of pain, functional/symptom status, hand-finger strength, median nerve ultrasonography measurements.

Patients who were evaluated by detailed clinical examination and medical history according to the inclusion and exclusion criteria were given written informed consent and assigned to one of the three treatment groups using block randomization. Basic sociodemographic information (age, gender, body mass index, employment status, education level, marital status,etc) and clinical data (dominant hand, duration of symptoms, comorbidities, hand to be treated, Tinel/Phalen sign, pain intensity, baseline electrophysiological parameters) will be recorded. The first group will consist of patients who have received peloid therapy at 45 degrees for a total of 15 sessions of 20 minutes, 5 days a week for 3 weeks with a home-based exercise program. The second group is a program consisting of adults who receive a total of 15 sessions of 20 minutes, paraffin bath treatment and home exercise program, 5 days a week for 3 weeks. Patients who only received home-based exercise program will be included in the 3rd group. During the treatment period, patients will be allowed to take only paracetamol for pain, if necessary, except for the medications they use continuously for comorbid reasons.

All groups were evaluated by a blinded assessor based on examination findings (Tinel/Phalen tests), pain intensity (VAS), hand grip strength (HGS), finger pinch strength (FGS), the Turkish version of the Boston Carpal Tunnel Questionnaire, the 4-Question Neuropathic Pain Questionnaire (DN4),Quick DASH Score, and ultrasound measurements (median nerve cross-sectional areas [CSA]) at the proximal insertion of the carpal tunnel (at the level of the scaphoid and pisiform bones and the distal wrist crease), both after treatment (three weeks/W3) and at three months post-treatment (W12).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Agreeing to participate voluntarily in the study
* Being diagnosed with mild or moderate idiopathic chronic CTS as a result of anamnesis, clinical examination and nerve conduction study

Exclusion Criteria:

* Presence of predisposing etiological factors for CTS such as diabetes mellitus, chronic kidney and liver disease, acromegaly, rheumatological diseases, acute trauma, hypothyroidism, etc.
* Being diagnosed with severe CTS
* Having a history of previous wrist surgery or trauma
* Having atrophy in the thenar region or weakness in the thenar muscles
* Having cervical radiculopathy, thoracic outlet syndrome, polyneuropathy, brachial neuropathy or proximal median nerve neuropathy
* Having had steroid injections in the last 3 months and taking oral steroid medications
* Being pregnant
* Having an open wound or rash in the wrist and its surroundings that would prevent treatment
* Patients who are receiving or will receive another/additional treatment for CTS
* Patients with a bifid median nerve, persistent median artery, ganglion cyst, tenosynovitis, or tendinitis in the wrist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
VAS pain | baseline, week 3 and week 12
  A 10 cm long line is drawn, this line is divided into 10 intervals of 10 mm width, 0: no pain and 10: the most severe pain is explained, and the patient is asked to mark the value corresponding to the resting pain and the pain during movement on the scale.
The Boston Carpal Tunnel Syndrome Questionnaire | baseline, week 3 and week 12
  The Turkish version of the Boston Carpal Tunnel Questionnaire score. It is used to evaluate the symptom severity and functionality of the patients. BCTQ is a questionnaire consisting of 2 parts: symptom severity scale (SSS) and functional status scale (FSS). Each item in both sections has 5 different answers that score between 1 and 5. The mean score is obtained by dividing the total score by the number of questions and ranges from 1 to 5, with a higher score indicating severe symptom.

SECONDARY OUTCOMES:
Hand grip strength | baseline, week 3 and week 12
  Following the definitions outlined in the literature, HGS will be measured using Jamar hand dynamometers. The patients will be asked to squeeze the dynamometer three times with maximum strength, allowing 30-60 seconds of rest between each attempt. The average force (in pounds/kg) will then be recorded.
Finger pinch strength | baseline, week 3 and week 12
  Following the definitions outlined in the literature, FGS will be measured using Baseline pinch dynamometers. The patients will be asked to squeeze the dynamometer three times with maximum strength, allowing 30-60 seconds of rest between each attempt. The average force (in pounds/kg) will then be recorded.
Douleur Neuropathique 4 | baseline, week 3 and week 12
  The DN4 is a short and simple screening test designed to help distinguish neuropathic pain from other types of pain, such as nociceptive pain. Neuropathic pain is assessed with four questions. The first two questions are based on the patient interview and the other two questions are based on the clinical examination.
Quick DASH Score | baseline, week 3 and week 12
  The purpose of the QuickDASH is to use 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The QuickDASH is a widely used reference of self-reported disability.
Ultrasonographic evaluation of the median nerve | baseline, week 3 and week 12
  Ultrasonographic evaluation of the median nerve will be performed with a LA2-14A transducer /superficial linear probe (Samsung). The cross-sectional areas (CSA) of the median nerve at the proximal inlet of the carpal tunnel will be recorded. To identify the entrance of the carpal tunnel, measurements will be taken at the level of the distal wrist crease, at the scaphoid and pisiform bones. The assessments were conducted with the patients seated, facing the clinician, with their elbow bent at approximately 90˚, forearm in a supine position, and fingers in a semiflexed posture. Measurements were obtained using the manual tracing feature of the ultrasound device, excluding the hyperechoic nerve sheathThe CSA (mm2) will be determined. The average of the three measurements will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No